CLINICAL TRIAL: NCT06648005
Title: Effect of Spinal Manipulative Therapy Combined with Brace in Moderate-severe Grade Adolescent Idiopathic Scoliosis: a Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Zhejiang Chinese Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-K-380-01
Record Dates: First submitted 2024-09-21; First posted 2024-10-18 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-08

CONDITIONS: Adolescent Idiopathic Scoliosis; Brace; Spinal Manipulative Therapy
Keywords: spinal manipulative therapye; brace; adolescent idiopathic scoliosis; moderate-grade; severe-grade; spinal deformity; quality of life
MeSH Terms: interventions — Braces

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SMTB group (Experimental): subjects in SMTB group and Brace group were all prescribed a brace with reference to the 2016 SOSORT guidelines and received preliminary assessment for brace design and fabrication at their first visit . Subjects were requested to wear orthosis 23 hrs/d and 1 hr for personal hygiene and exercise activities . The subjects were treated for 12 months . In addition, interview for compliance was launched when the subjects came to the scoliosis clinic for follow-up visits.
  Besides bracing, the SMTB group was treated with spinal manipulative therapy . If discomfort occurs, we will stop the treatment immediately. Spinal manipulation is performed twice a week. Two doctors with 10 years of clinical experience will perform all examinations and manipulations. Intensive training was given to the physiotherapists in spinal manipulation. The doctors took the medical history of all participants and performed a clinical examination.
  Interventions: Procedure: the spinal manipulative therapy combined brace
- Brace group (Active Comparator): Upon enrollment, subjects in SMTB group and Brace group were all prescribed a brace with reference to the 2016 SOSORT guidelines and received preliminary assessment for brace design and fabrication at their first visit. Subjects were requested to wear orthosis 23 hrs/d and 1 hr for personal hygiene and exercise activities. The subjects were treated for 12 months. In addition, interview for compliance was launched when the subjects came to the scoliosis clinic for follow-up visits.
  Interventions: Other: brace

INTERVENTIONS:
Procedure: the spinal manipulative therapy combined brace — Besides bracing, the SMTB group was treated with spinal manipulative therapy. If discomfort occurs, we will stop the treatment immediately. Spinal manipulation is performed twice a week. Two doctors with 10 years of clinical experience will perform all examinations and manipulations. Intensive training was given to the physiotherapists in spinal manipulation. The doctors took the medical history of all participants and performed a clinical examination.
  Arms: SMTB group
Other: brace — Subjects were requested to wear orthosis 23 hrs/d and 1 hr for personal hygiene and exercise activities. The subjects were treated for 12 months. In addition, interview for compliance was launched when the subjects came to the scoliosis clinic for follow-up visits.
  Arms: Brace group

SUMMARY:
Objective: To determine whether spinal manipulative therapy combined with brace is superior to a control of brace alone in improving spinal deformity and quality of life of moderate-severe grade AIS.

Design: It is a prospective randomized controlled study. Patients who met the inclusion criteria were randomly assigned to either the spinal manipulative therapy combined brace group (SMTB) or the Brace group. All participants were prescribed with a GBW brace and the spinal manipulative regimen was provided to the subjects in the SMBT group. Cobb angle, angle of trunk rotation (ATR), quality of life (SRS-22), progression rates and surgical rates of the subjects were measured at baseline to the 12-month follow-up.

DETAILED DESCRIPTION:
Introduction Adolescent idiopathic scoliosis (AIS) is a complex three-dimensional deformity of the spine that primarily affects children and adolescents. It is characterized by coronal scoliosis, sagittal imbalance, and horizontal rotation of the spine. The global prevalence of AIS is estimated to be around 2-3%, with a higher proportion of female patients. Moderate-severe grade AIS may lead to physical deformities including razorback, shoulder imbalance and chest deformity, and even affect cardiopulmonary function and irreversible damage to nerves. In addition, patients with AIS are often associated with moderate to severe psychological disorders. Research has confirmed that if left untreated, approximately 60% of individuals with moderate-severe AIS will experience progression of their scoliosis. Moreover, about 30% moderate-severe AIS will suffer from physical deformities, chronic pain, and psychosocial disorders, such as anxiety and depression, during adulthood.

AIS is classified into three categories based on the extent of spinal curvature, measured by the Cobb angle: mild (<20°), moderate (20-40°), and severe (>40°). Current guidelines, such as the 2016 SOSORT guidelines [8], recommend the primary treatment regimen for moderate AIS to consist of bracing therapy and rehabilitative exercises. This regimen aims to reduce pain, improve posture, and control further progression of scoliosis, ultimately aiming to avoid surgery. However, in clinical practice, prolonged bracing alone can have negative impacts on growth and development, including pressure sores, back pain, decreased respiratory function and potential mental health issues.

It is now generally accepted that severe-grade AIS with skeletally immature need to undergo surgical corrective surgery. But this approach involves relatively high-cost issues and risk of complications due to the invasive, complex nature of the procedure. As a result of these problems, some patients with AIS who are considered to be surgical candidates, as well as their parents, expressly resist surgery and seek more aggressive conservative treatment. In recent years, more and more reports in the literature have shown that conservative treatment still has a certain therapeutic effect on AIS >40° (35%-91%).But this efficacy is affected by a number of risk factors. There is still a need to explore an active conservative treatment for AIS, aims to correct scoliosis, avoid surgery.

Spinal manipulative therapy (SMT), as a complementary and alternative therapy for AIS, is a skilled hand manipulative technique, including massage, chiropractic, osteopathy, and Tuina (traditional Chinese manipulation). Extensive research has demonstrated its effectiveness in reducing pain, decreasing scoliosis angle and improving overall quality of life in patients with AIS. Our team has also observed the corrective effect of SMT on moderate-grade AIS in the clinic beforehand.

However, what needs to be acknowledged is that existing research on the efficacy of SMT for AIS is hampered by the heterogeneity of clinical research protocols and the lack of high-quality randomized controlled trials (RCTs). To ensure consistency in the application of SMT and to obtain more reliable evidence of its efficacy in the clinical management of AIS, our team conducted this RCT to observe the effect of SMT on improving spinal deformity and quality of life in patients with moderate-severe AIS.

Methods Trial design This study employed a randomized controlled clinical trial design, employing a 1:1 allocation ratio to assign participants either to the intervention group receiving spinal manipulative therapy combined with brace (SMTB) or the control group receiving brace. Patient enrollment commenced in January 2022, and follow-up treatment concluded in December 2023. The study strictly adhered to the CONSORT guidelines, and ethical approval was obtained from the Ethics Committee of the First Hospital Affiliated to Zhejiang University of Traditional Chinese Medicine (2022-K-380-01). Furthermore, the study protocol was registered with ClinicalTrials.gov (ChiCTR2200057023).

Participants The participants who fulfilled the subject selection criteria were all enrolled from Scoliosis Treatment Centre of The First Affiliated Hospital of Zhejiang Chinese Medical University. The target population for this study was those with moderate-severe grade AIS who met the comprehensive inclusion criteria recommended by the Scoliosis Research Society (SRS) and the Society on Scoliosis Orthopedic and Rehabilitation Treatment (SOSORT): (1) 10-18 years old; (2) primary curve magnitude 20°-60° Cobb angle; (3) signing informed consent and cooperating with treatment and follow-ups. The subjects with neuromuscular, rheumatic, cardiovascular, pulmonary, congenital spine-related disorders, psychiatric problems, or a history of spinal surgery were excluded from the study.

Intervention Upon enrollment, subjects in SMTB group and Brace group were all prescribed a brace with reference to the 2016 SOSORT guidelines and received preliminary assessment for brace design and fabrication at their first visit. Subjects were requested to wear orthosis 23 hrs/d and 1 hr for personal hygiene and exercise activities. The subjects were treated for 12 months. In addition, interview for compliance was launched when the subjects came to the scoliosis clinic for follow-up visits.

Besides bracing, the SMTB group was treated with spinal manipulative therapy. If discomfort occurs, the investigators will stop the treatment immediately. Spinal manipulation is performed twice a week. Two doctors with 10 years of clinical experience will perform all examinations and manipulations. Intensive training was given to the physiotherapists in spinal manipulation. The doctors took the medical history of all participants and performed a clinical examination.

1. Finger-pressing manipulation. Subjects were kept in the prone position. Continuous pressure is applied to the treated section using manipulator's own thumb to relax the thoracic vertebra concave side muscle groups. It takes 5 minutes(Figure 1 finger-pressing manipulation.).
2. Elbow-pressing manipulation. Subjects were kept in the prone position. Continuous pressure is applied to the treated section using manipulator's elbow to relax the lumbar vertebra concave side muscle groups. It takes 5 minutes(Figure 2 Elbow-pressing manipulation.).
3. Thoracic vertebra pulling manipulation. Take the left thoracic curve as an example. The patient was placed in a sitting position with his left hand resting on his neck and his left elbow bent. The operator's left hand was passed through the patient's left elbow and placed on top of the patient's left hand, with the right hand gripping the patient's left upper arm. The operator's right hand was pulled upward for pulling the thoracic vertebrae, sometimes with localized joint popping.(Figure 3 Thoracic vertebra pulling manipulation.).
4. Lumbar oblique-rotation- pulling manipulation. Take the left lumbar curve as an example. The patient was placed in the left lateral decubitus position. The surgeon stands to the left of the patient. The right hand was placed on the right shoulder of the patient to fix the right shoulder. The left hand was placed on the patient's right pelvis for fixation. The surgeon rotated the patient's lumbar spine to its maximum. The left hand is rotated ventrally and pulled down to create a momentary force, sometimes with localized joint popping.( Figure 4. Lumbar oblique-rotation- pulling manipulation).

Compliance supervision To promote subject cooperation, the subjects and their parents will be educated before treatment about the risk of progression of scoliosis, its harmfulness, and the necessity for treatment. When a subject's compliance begins to falter, their parents will be encouraged to encourage the subjects to continue training.

Outcomes General patient characteristics collected at baseline included age(y), sex(female, male), weight(kg), height(cm), body mass index (BMI,kg/m2), risser grade, and location of the major curve(thoracic, thoracolumbar, lumbar). Assessments were performed at baseline and after 3, 6, 12 months of treatment for each patient. The final measurements were taken 24 hours after removal of the brace. Cobb angle, trunk rotation angle (ATR), and quality of life of the participants were assessed by the same researcher who conducted the interviews.

Body mass index (BMI) is a statistical index using a person's weight and height to provide an estimate of body fat in males and females of any age. It is calculated by taking a person's weight, in kilograms, divided by their height, in meters squared, or BMI = weight (in kg)/ height^2 (in m^2). The number generated from this equation is then the individual's BMI number.

Risser grade is a staging system of bone maturity based on the ossification of the iliac apophysis, ranging from 0 to 5, with higher grades indicating Greater maturity.

Location of the major curve judgement according to the location of the apex: thoracic (apex between T2 and T11), thoracolumbar (apex in T12 or L1), and lumbar (apex between L2 and L4).

The primary outcome measure was the curve reduction of 6° or more (treatment success) or curve reduction of less than 6° seen on pretherapy and post-treatment posteroanterior standing radiographs compared with the inclusion radiograph (treatment failure).

Radiographic measurements were conducted through radiographic images in the Digital Imaging and Communications in Medicine image format using the picture archiving and communication system, version 23.1 clinical imaging tool (Sectra PACS).

A range of secondary outcomes were measured which was scoliosis related： Cobb angle is the gold standard for evaluating the degree of scoliosis. Measurement of Cobb angle was carried out at baseline and after 12-month of treatment, and changes in its degree were observed to determine whether the scoliosis had improved or progressed.

ATR was measured using the Bunnell's sociometer in a standing forward flexed position, which is considered to be sensitive, specific, and reliable. The greater the angle, the more pronounced the razorback, and the worse the subject's posture. The ATR was collected at baseline and after 3, 6, 12month of treatment.

The Scoliosis Research Society-22 (SRS-22) questionnaire, used to assess health-related quality of life, is a simple yet practical questionnaire currently available for AIS, with good validity and retest reliability for clinical application. It consists of five dimensions: function, pain, self-image, mental health (five questions each) and satisfaction with treatment (two questions), for a total of 22 questions, each rated from 1 (worst) to 5 (best). The higher the score, the better the subject's quality of life. This questionnaire was assessed at subject enrollment and after 6, 12month of treatment.

Randomization and Blinding A random number sequence was generated by SPSS Statistics, version 23.0 (IBM Corp) and used to completely randomize the included all patients into groups. They were divided into intervention and control groups. The grouping information was made into a randomization card and kept in sequentially numbered and opaque envelopes. The doctor in charge of treatment opened the envelopes to obtain the grouping code according to the order in which the patients were enrolled. Due to the specificity of the manipulation, this study could not be blinded to subjects and clinicians, but researchers who assessed efficacy and analyzed the data were blinded to treatment assignment.

Safety monitoring and adverse events All expected or unexpected adverse events from this study will be recorded and monitored. Patients suffered from any adverse events related to this study will also receive free treatment. There will be a fast channel for the emergency or abnormal sensations requiring the clinician's intervention.

Statistical analysis When calculating the sample size, the response rate was taken as the primary indicator for assessing the efficacy of manipulation in patients who with AIS. Based on data from and the pre-test results, the control group effectiveness was 68.0%, whereas it was anticipated that the treatment group effectiveness would achieve 89.5%. By utilizing the PASS software version 15 and setting an alpha level of 0.05 and power (1-β) of 0.80, it was determined that a minimum of 106 subjects per group was necessary. Taking into account 12 months of continuous treatment and potential losses, it was ultimately decided to include 118 subjects per group.

All primary analyses were conducted according to the intention-to-treat principle. The investigators did efficacy analyses in the full analysis set and per protocol set, which included all randomized patients who received at least one session of treatment and had at least one efficacy measure.The primary analysis population included all patients with Cobb angle data reported within the time window defined in the protocol (-4 week to 0 weeks around the 12-month post-randomization follow-up timepoint). A sensitivity analysis was performed comparing the intention to treat analysis data against per-protocol data exclusively from patients who complied with the study protocol.

The investigators did safety analyses in the safety set, which included all randomized patients who received at least one session of spinal manipulative therapy or brace.

All statistical analyses were performed using SPSS statistics, version 23.0 (IBM Corp). Continuous and discrete parameters were measured using parametric or nonparametric tests for group comparisons. The Shapiro-Wilks test was used to test the normality of each study parameter. Independent t-test was used for comparison between groups and paired t-test for comparison within groups. Meanwhile, the chi-square test was used for comparison between groups for count data. The statistical significance level was set at P<0.05.

All statistical analyses of the primary outcome were conducted by 2 independent statisticians, who were blinded to intervention and assigned to each patient participating in the study.

Patient and public involvement No patients were involved in the design or conduct of the study, in setting the research question, or in determining the outcome measures of this study, nor did they have any input on data analysis, interpretation, or writing up of results.

ELIGIBILITY:
The target population for this study was those with moderate-severe grade AIS who met the comprehensive inclusion criteria recommended by the Scoliosis Research Society (SRS) and the Society on Scoliosis Orthopedic and Rehabilitation Treatment (SOSORT).

Inclusion Criteria:

1. 10-18 years old
2. Primary curve magnitude 20°-60° Cobb angle
3. Signing informed consent and cooperating with treatment and follow-ups

Exclusion Criteria:

1. The subjects with neuromuscular, rheumatic, cardiovascular, pulmonary, congenital spine-related disorders
2. Psychiatric problems
3. A history of spinal surgery

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 169 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
curve reduction | Assessments were performed at baseline and after 3, 6, 12 months of treatment for each patient
  the curve reduction of 6° or more (treatment success) or curve reduction of less than 6° seen on pretherapy and post-treatment posteroanterior standing radiographs compared with the inclusion radiograph (treatment failure) .
  Radiographic measurements were conducted through radiographic images in the Digital Imaging and Communications in Medicine image format using the picture archiving and communication system, version 23.1 clinical imaging tool (Sectra PACS).

SECONDARY OUTCOMES:
Cobb angle | at baseline and after 12-month of treatment
  Cobb angle is the gold standard for evaluating the degree of scoliosis. Measurement of Cobb angle was carried out at baseline and after 12-month of treatment, and changes in its degree were observed to determine whether the scoliosis had improved or progressed.
ATR | The ATR was collected at baseline and after 3, 6, 12month of treatment
  ATR was measured using the Bunnell's sociometer in a standing forward flexed position, which is considered to be sensitive, specific, and reliable. The greater the angle, the more pronounced the razorback, and the worse the subject posture.
The Scoliosis Research Society-22 (SRS-22) questionnaire | This questionnaire was assessed at subject enrollment and after 6, 12month of treatment
  The Scoliosis Research Society-22 (SRS-22) questionnaire, used to assess health-related quality of life, is a simple yet practical questionnaire currently available for AIS, with good validity and retest reliability for clinical application. It consists of five dimensions: function, pain, self-image, mental health (five questions each) and satisfaction with treatment (two questions), for a total of 22 questions, each rated from 1 (worst) to 5 (best). The higher the score, the better the subject's quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Zhejiang Chinese Medical University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu C, Wu YQ, Wang KQ, Wen Y, Li QS, Chen XM, Tang D, Du HG, Chen S. Spinal Manipulative Therapy for Moderate-to-Severe Adolescent Idiopathic Scoliosis: A Randomized Controlled Trial. Chin J Integr Med. 2025 Dec 22. doi: 10.1007/s11655-025-4228-8. Online ahead of print. PMID 41428026